CLINICAL TRIAL: NCT02782975
Title: A Randomized, Open-Label, Parallel-Arm Study to Assess the Absolute Bioavailability of a Single, Fixed Subcutaneous Dose of Aducanumab (BIIB037) in Healthy Subjects Compared to a Single, Weight-Based Intravenous Dose
Brief Title: Absolute Bioavailability of a Single, Fixed Subcutaneous Dose of Aducanumab in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 221HV102
Record Dates: First submitted 2016-05-23; First posted 2016-05-26 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — aducanumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- aducanumab IV (Experimental): Infusion of aducanumab over approximately 1 hour
  Interventions: Drug: aducanumab
- aducanumab SC (Experimental): Subcutaneously via injection
  Interventions: Drug: aducanumab

INTERVENTIONS:
Drug: aducanumab
  Other Names: BIIB037

SUMMARY:
The primary objectives of this study are to evaluate the absolute bioavailability of a single, fixed sub-cutaneous (SC) dose of aducanumab compared with a single, weight-based intra-venous (IV) dose in healthy participants and to characterize the pharmacokinetics (PK) profile of aducanumab. The secondary objectives are to evaluate the safety and tolerability of aducanumab administered via SC and IV routes in healthy participants and to characterize additional PK parameters of a single, fixed SC dose of aducanumab and a weight-based IV dose in healthy participants.

ELIGIBILITY:
Key Inclusion Criteria:

* A minimum weight of 45 kg, inclusive, at Day -1.
* All women of childbearing potential and all men must practice highly effective contraception during the study and be willing and able to continue contraception for 24 weeks after study treatment dosing (Day 1).
* Must be in good health (as determined by the Investigator) based on the medical history and screening evaluations.

Key Exclusion Criteria:

* Mini mental state examination (MMSE) score of <27 at Screening.
* History of any clinically significant cardiac, endocrinologic, hematologic, hepatic, gastrointestinal, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, or renal disease, or other major disease, as determined by the Investigator.
* History of severe allergic or anaphylactic reactions that in the opinion of the Investigator is likely to be exacerbated by any component of the study treatment.
* History of malignant disease, including solid tumors and hematologic malignancies (with the exception of basal cell and squamous cell carcinomas of the skin that have been completely excised prior to study entry).
* History of, or positive test result at Screening for, human immunodeficiency virus (HIV).
* Positive test result at Screening for hepatitis C virus antibody (HCVAb).
* Positive test result at Screening for hepatitis B virus (defined as positive for both, hepatitis B surface antigen [HBsAg] AND hepatitis B core antibody [HBcAb]).
* Chronic, recurrent, or serious infection (e.g., pneumonia, septicemia) as determined by the Investigator, within 90 days prior to Day -1.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2016-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
PK parameter of SC dose of aducanumab: Absolute Bioavailability | 13 weeks
PK parameter of IV dose of aducanumab: Area under the concentration-time curve from time zero to infinity (AUCinf) | 13 weeks
PK parameter of SC dose of aducanumab: Area under the concentration-time curve from time zero to infinity (AUCinf) | 13 weeks
PK parameter of aducanumab: Maximum observed concentration (Cmax) | 13 weeks
PK parameter of SC route of aducanumab: Time to reach maximum observed concentration (Tmax) | 13 weeks

SECONDARY OUTCOMES:
Number of participants experiencing Adverse Events (AEs) and Serious Adverse Events (SAEs) | 13 weeks
Number of participants with clinically significant vital sign abnormalities | 13 weeks
Number of participants with clinically significant laboratory assessment abnormalities | 13 weeks
Number of participants with clinically significant 12-lead electrocardiograms (ECGs) abnormalities | 13 weeks
PK parameter of aducanumab: Area under the concentration-time curve from time zero to the time of the last measurable sample (AUClast) | 13 weeks
PK parameter of aducanumab: Terminal elimination half-life (t1/2) | 13 weeks
PK parameter of aducanumab: Volume of distribution (Vd) | 13 weeks
PK parameter of aducanumab: Apparent total body clearance (CL/F) | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (2):
- United States (2):
  - Research Site, Evansville, Indiana
  - Research Site, Dallas, Texas